CLINICAL TRIAL: NCT01003340
Title: A Randomized Controlled Trial of a Community Health Worker Home-Based Asthma Intervention
Brief Title: A Community Health Worker Home Intervention to Improve Pediatric Asthma Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: American Lung Association (Other)
Responsible Party: Principal Investigator, Marina Reznik, principal investigator, Montefiore Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 07-10-360; CG-120837-N (Other Grant/Funding Number: American Lung Association)
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Asthma
Keywords: asthma; children; community health workers; home intervention
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Wee Wheezers asthma education (Experimental): 6 lesson asthma education delivered at home by Community Health Workers
  Interventions: Behavioral: Wee Wheezers

INTERVENTIONS:
Behavioral: Wee Wheezers — The intervention, Wee Wheezers, modified to the needs of the targeted population will include 6 bi-weekly 1 hour educational home visits conducted by Community Health Workers at homes of children with persistent asthma
  Other Names: Wee Wheezers at Home

SUMMARY:
The investigators propose to test the hypothesis that a home-based asthma intervention, the Wee Wheezers program, delivered by the Community Health Workers and tailored to the needs of the investigators community, will improve anti-inflammatory medication adherence, parental asthma knowledge and management behaviors, which in turn will reduce asthma morbidity (defined as days with asthma symptoms) and health care utilization (defined as asthma-related Emergency Department visits) among low-income, minority children with persistent asthma in the Bronx.

DETAILED DESCRIPTION:
Asthma disproportionately burdens low-income inner city and minority children residing in inner cities. Daily use of inhaled corticosteroids (ICS) control symptoms and reduce asthma morbidity. Less then 50% of children with persistent asthma adhere to such therapy. Poor adherence to ICS medications is one of the major contributors to asthma morbidity. One way to reduce asthma disparities is to work in partnership with communities. Community Health Workers (CHWs) share the ethnic, cultural, social, and environmental experiences of the people in the community. Although, CHW home interventions have been successful in reducing asthma allergens, no studies using CHWs to deliver a previously identified evidence-based home intervention to improve ICS adherence and health outcomes in a population of inner-city, minority children with persistent asthma have been found. Objective: To evaluate the effectiveness of an evidence-based asthma home intervention, the Wee Wheezers program, tailored to the needs of the community and delivered by CHWs, in improving medication adherence, health outcomes and parental management behaviors among low-income, minority children with persistent asthma in the Bronx.

ELIGIBILITY:
Inclusion Criteria:

* children 2-9 years of age with persistent asthma
* children being currently prescribed ICS in the Metered Dose Inhaler (MDI) form
* if the child is 2 years of age at the time of the recruitment, he/she must have at least two prior episodes of wheezing treated and reversible with beta-agonists
* primary caregiver speaks English or Spanish
* family has a phone.

Exclusion Criteria:

* children with other chronic pulmonary diseases (e.g, cystic fibrosis, bronchopulmonary dysplasia) or presence of tracheostomy

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 188 (Actual)
Dates: Start 2009-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
mean number of asthma symptom days | baseline and every 8 weeks during the 12-months study period
  average of asthma symptom days

SECONDARY OUTCOMES:
adherence to Inhaled Corticosteroid | baseline, 4 weeks, 8 weeks, and 12 weeks after beginning of intervention
  survey evaluating medication adherence
asthma-related Emergency Department visits | baseline, 3-, 6- and 12-months follow-up
  number of ED visits
parental asthma knowledge and management behaviors | baseline, 3-, 6- and 12-months follow-up
  survey evaluating asthma knowledge and management behavior

CONTACTS AND LOCATIONS:
Overall Officials: Marina Reznik, MD, MS, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Group- CHCC, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reznik M, Ozuah PO. Measurement of inhaled corticosteroid adherence in inner-city, minority children with persistent asthma by parental report and integrated dose counter. J Allergy (Cairo). 2012;2012:570850. doi: 10.1155/2012/570850. Epub 2012 Mar 15. PMID 22505947
- [Result] Reznik M, Silver EJ, Cao Y. Evaluation of MDI-spacer utilization and technique in caregivers of urban minority children with persistent asthma. J Asthma. 2014 Mar;51(2):149-54. doi: 10.3109/02770903.2013.854379. Epub 2013 Oct 22. PMID 24131031
- [Result] Reznik M, Jaramillo Y, Wylie-Rosett J. Demonstrating and assessing metered-dose inhaler-spacer technique: pediatric care providers' self-reported practices and perceived barriers. Clin Pediatr (Phila). 2014 Mar;53(3):270-6. doi: 10.1177/0009922813512521. Epub 2013 Dec 12. PMID 24336438